CLINICAL TRIAL: NCT04275583
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance and Pharmacokinetics of TQB3602 Capsule
Brief Title: A Study to Evaluate the Tolerance and Pharmacokinetics of TQB3602 Capsule
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3602-I-01
Record Dates: First submitted 2020-02-16; First posted 2020-02-19 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3602 capsule (Experimental): TQB3602 capsule administered orally on day 1, 8, 15 in 28-day cycle.
  Interventions: Drug: TQB3602

INTERVENTIONS:
Drug: TQB3602 — This is a kind of proteasome inhibitor.

SUMMARY:
This is a study to evaluate the tolerance, dose-limiting toxicity (DLT), phase II recommended dose (RP2D), and maximum tolerated dose (MTD) of single and multiple oral doses of TQB3474 in patients with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1.Understood and signed an informed consent form. 2.18 and 75 years old , male or female. 3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2.

  4. Life expectancy ≥12 weeks. 5. Relapsed/refractory multiple myeloma had received at least two treatment methods.

  6. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

Exclusion Criteria:

* 1. Hypersensitivity to TQB3602 or its excipient. 2. Has peripheral nerve diseases ≥ grade 2. 3. Has diarrhea grade > 1 during screening period. 4. Has received chemotherapy, radiotherapy, targeted therapy, immunotherapy, or other systemic antitumor therapies within 14 days before the first dose.

  5. Has received ixazomib and less than 5 half-life before the first dose. 6. Has received allogeneic stem cell transplant. 7. Pregnant or lactating women. 8. Has participated in other clinical trials within 4 weeks before participating in this trial.

  9. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days
  Subjects appear the following toxic reaction relate to the drug after treatment within 28 days ：III °or above of non-hematological toxicity, IV° hematological toxicity , III ° neutropenia associated with fever, III ° thrombocytopenia with bleeding.

SECONDARY OUTCOMES:
Cmax | 0hour, 15minutes, 0.5hour, 1hour, 1.5hour, 2hour, 4hour, 8hour, 12hour, 24hour, 48hour, 96hour, 120hour, 144hour after oral administration of day 1 and day 15; Hour 0 of day 8 , hour 0 of day 29.
  Cmax is the maximum plasma concentration of TQB3602 or metabolite(s).
Tmax | 0hour, 15minutes, 0.5hour, 1hour, 1.5hour, 2hour, 4hour, 8hour, 12hour, 24hour, 48hour, 96hour, 120hour, 144hour after oral administration of day 1 and day 15; Hour 0 of day 8 , hour 0 of day 29.
  To characterize the pharmacokinetics of TQB3602 by assessment of time to reach maximum plasma concentration.
AUC0-t | 0hour, 15minutes, 0.5hour, 1hour, 1.5hour, 2hour, 4hour, 8hour, 12hour, 24hour, 48hour, 96hour, 120hour, 144hour after oral administration of day 1 and day 15; Hour 0 of day 8 , hour 0 of day 29.
  To characterize the pharmacokinetics of TQB3602 by assessment of area under the plasma concentration time curve from zero to infinity.

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital, Sichuan University, Chengdu, Sichuan, China